CLINICAL TRIAL: NCT04631991
Title: Association Between Retinal Microvasculature and Optic Disc Alterations in Non-pathological High Myopia With Optical Coherence Tomography Angiography
Brief Title: Association Between Retinal Microvasculature and Optic Disc Alterations in Non-pathological High Myopia With OCTA
Status: Completed | Type: Observational
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Aslı Çetinkaya Yaprak, Principal Investigator, Akdeniz University
Other Study IDs: 18062020-167
Record Dates: First submitted 2020-11-11; First posted 2020-11-17 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-pathological high myopia: Comprehensive ophthalmologic examination
  Interventions: Diagnostic Test: Comprehensive ophthalmologic examination
- Control: Comprehensive ophthalmologic examination
  Interventions: Diagnostic Test: Comprehensive ophthalmologic examination

INTERVENTIONS:
Diagnostic Test: Comprehensive ophthalmologic examination — Measurements of best-corrected visual acuity, refractive error, intraocular pressure, axial length, slit lamp examination of the anterior segment, dilated fundus examination, and optical coherence tomography angiography imaging.

SUMMARY:
Non-pathological high myopia patients and controls undergoing a comprehensive ophthalmologic examination are included. The Optical Coherence Tomography Angiography (OCTA) software automatically segments these full-thickness retinal scans into the superficial and deep inner retinal vascular plexuses, outer retina, and choriocapillaris (CC). The vascular density in the superficial and deep retinal vascular zones is calculated automatically by the software, and the foveal avascular zone (FAZ) and foveal density (FD) are also automatically determined. Choroidal thickness is calculated manually by two retinal specialists, and the average value was used.

DETAILED DESCRIPTION:
Non-pathological high myopia patients and controls undergoing a comprehensive ophthalmologic examination, including measurements of best-corrected visual acuity, refractive error; intraocular pressure, axial length, slit lamp examination of the anterior segment, dilated fundus examination and OCTA imaging are included. The best-corrected visual acuity is convert into the logarithm of minimal angle resolution. The OCTA images are independently graded and assessed by two retinal specialists. The software automatically segmented these full-thickness retinal scans into the superficial and deep inner retinal vascular plexuses, outer retina, and choriocapillaris (CC). The vascular density in the superficial and deep retinal vascular zones is calculated automatically by the software, and the foveal avascular zone (FAZ) and foveal density (FD) are also automatically determined. Choroidal thickness is calculated manually by two retinal specialists, and the average value was used.

Right eye of each participant is included in the study. If the right eye shows any exclusion criteria, then the left eye is selected for enrollment. Eyes with an AL longer than 26 mm are included in the HM group. The classification of myopic maculopathy is applied in identification of fundus alterations. Patients with category 0 (no myopic retinopathy lesions) and category 1 (tessellated fundus) are included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with category 0 (no myopic retinopathy lesions)
* Patients with category 1 (tessellated fundus)

Exclusion Criteria:

* poor image quality (signal strength index (SSI) <60) due to unstable fixation
* IOP >21 mm Hg; logMAR > 0.1
* pre-existing ophthalmic pathologies
* prior ocular surgery
* systemic chronic disease which can cause retinopathy
* such as diabetes mellitus, hypertension etc.

Ages: 18 Years to 50 Years | Sex: All
Age Groups: Adult
Study Population: Study population includes a convenience sampling from the patients admitted to outpatient clinic between November 2020 and December 2020.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-11-10 (Actual); Primary Completion 2020-12-05 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Optic nerve head vessel density | 10 minutes
  Optic nerve head vessel density assessed with optical coherence tomography angiography

SECONDARY OUTCOMES:
Choriocapillaris flow area | 10 minutes
  Choriocapillaris flow area assessed with optical coherence tomography angiography
Subfoveal choroidal thickness | 10 minutes
  Subfoveal choroidal thickness assessed with optical coherence tomography angiography
Foveal avascular zone | 10 minutes
  Foveal avascular zone assessed with optical coherence tomography angiography
Subfoveal central macular thickness | 10 minutes
  Subfoveal central macular thickness assessed with optical coherence tomography angiography

CONTACTS AND LOCATIONS:
Locations (1):
- Aslı Çentinkaya Yaprak, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yaprak AC, Yaprak L. Retinal microvasculature and optic disc alterations in non-pathological high myopia with optical coherence tomography angiography. Graefes Arch Clin Exp Ophthalmol. 2021 Nov;259(11):3221-3227. doi: 10.1007/s00417-021-05216-x. Epub 2021 May 7. PMID 33961111